CLINICAL TRIAL: NCT00538044
Title: the Clinical Research Using Simvastatin as a Medication to Treat Advanced Secondary Pulmonary Hypertension
Brief Title: Simvatstatin Used to Treat Pulmonary Hypertension
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gan1; Anzhen1
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary hypertension; simvastatin; advanced pulmonary hypertension secondary to congenital heart disease; advanced pulmonary hypertension secondary to chronic pulmonary embolism
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1simvastatin group (Experimental): before the operation, the patient start the simvastatin medication on the dosage of 40mg per day
  Interventions: Drug: simvastatin
- 2contral group (No Intervention): just do routin operation with no use of simvastatin, other medication is exact the same as the simvastatin group

INTERVENTIONS:
Drug: simvastatin — medication with simvastation on the dosage of 40mg per day before the operation and all the time after the operation
  Arms: 1simvastatin group

SUMMARY:
we try to use simvastatin in the treatment of advanced pulmoary hypertension secondary to congenital heart disease or chronic pulmonary embolism before and after the operation.

DETAILED DESCRIPTION:
advanced pulmonary hypertension is refractory to the medication in use nowaday, especially pulmonary hypertension secondary to congenital heart disease or chronic pulmonary embolism.It is revealed that statins may intefere the pathogenisis of the pulmonary hypertension in many key poing, such as improving apotosis or inhiting the proliferation of pulmonary vascular smooth muscle cell. so we try to use simvastatin in the treatment of advanced pulmoary hypertension secondary to congenital heart disease or chronic pulmonary embolism before and after the operation.

ELIGIBILITY:
Inclusion Criteria:

* pasp>50mmHg

Exclusion Criteria:

* pasp<50mmhg

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2009-01; Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
the simvastatin can alleviate pulmonary hypertension
pulmonary pressure

SECONDARY OUTCOMES:
simvastatin can highten the perioperative and long term survaval rate and the living quality

CONTACTS AND LOCATIONS:
Overall Officials: Huili Gan, MD,Ph.D., Study Chair — Beijing Anzehn Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China